CLINICAL TRIAL: NCT02694458
Title: Comparison of Two Dosage Adjustment Strategies of Vancomycin in Children
Acronym: OPTIBAYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A01545-44
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Methicillin-resistant Staphylococcal Infections
Keywords: Vancomycin; Children; Infection; Antibiotic; Methicillin-resistant Staphylococcus aureus (MRSA); Population-based pharmacokinetic modeling; Pharmacokinetics; Pharmacodynamics; Bayesian approach; Therapeutic drug monitoring
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modeling arm (Experimental): Early vancomycin monitoring and bayesian dosage adjustment
  Interventions: Other: Early vancomycin monitoring and bayesian dosage adjustment
- Control arm (Sham Comparator): Usual vancomycin dose and monitoring strategy
  Interventions: Other: usual vancomycin dose and monitoring strategy

INTERVENTIONS:
Other: Early vancomycin monitoring and bayesian dosage adjustment — Measure of vancomycin serum concentration at the 3rd hour of treatment and adjustment of vancomycin dosage at the 6th hour of treatment using a bayesian approach. Then measure of vancomycin serum concentration at the 24th hour of treatment.
  Arms: Modeling arm
Other: usual vancomycin dose and monitoring strategy — Vancomycin serum concentration will be measured at the 24th hour of treatment.
  Arms: Control arm

SUMMARY:
Vancomycin is the standard first-line treatment for MRSA infections and a first-line empiric therapy. The relationship between exposure to vancomycin and efficacy is admitted but because of an important intersubject variability, therapeutic exposure isn't usually achieved.

The primary aim of this randomized controlled trial is to evaluate a new early dosage adjustment strategy of vancomycin in children, comparing it to the usual treatment strategy.

Using a bayesian approach, the purpose is to achieve earlier a therapeutic and non-toxic exposure to vancomycin.

The primary hypothesis is that an early dosage adjustment strategy using a bayesian approach will allow patients to achieve the vancomycin pharmacological target faster than with the usual treatment strategy.

DETAILED DESCRIPTION:
Introduction/ Clinical significance :

Staphylococcus aureus is a common cause of serious infections. Methicillin-resistant Staphylococcus aureus (MRSA) are one of the most common causes of nosocomial antibiotic resistant bacterial infections in the world. According to the last data from the European Antimicrobial Resistance Network, in 2014, 17,4 % of invasive staphylococcal infections are due to MRSA in France, with proportions of up to 56 % in some regions in the European Economic Area (EEA). In the United-States of America, MRSA reach 50 % of Staphylococcus isolates in some studies. Vancomycin is the standard first-line treatment for MRSA infections and a first-line empiric therapy.

To optimize good clinical outcomes for invasive MRSA infections using pharmacokinetics-pharmacodynamics of vancomycin, studies support targeting area under the curve (AUC) of the serum concentration versus time over 24 hours to minimum inhibitory concentration (MIC) ratio ≥ 400, which frequently correlates to a trough concentration of 15 - 20 mg/L when the MIC is 1 mg/L. Because of few consensus regarding the dosage to use and high intersubject variability, this pharmacological target is difficult to reach in children, which may lead to a delayed infection control and an increase of vancomycin toxicity-related side effects.

Aims :

The primary aim is to evaluate an early dosage adjustment strategy of vancomycin in children, comparing it to the usual treatment strategy.

Using a bayesian approach, the main purpose is to achieve earlier a therapeutic and non-toxic exposure to vancomycin.

The secondary aims are to compare with the usual treatment strategy 1) the proportion of subjects with vancomycin serum concentration within the concentration targets at the 24th hour of treatment, and 2) the clinical (in terms of fever), biological (in terms of CRP) and bacteriological (in terms of blood culture) efficacy of this early dosage adjustment strategy of vancomycin.

Hypothesis :

This study hypothesizes that early dosage adjustment strategy of vancomycin using a bayesian approach will be superior to usual treatment strategy in achieving the pharmacological target of vancomycin at the 24th hour of treatment in children.

Methodology :

As part of routine care, a prospective open-label randomized controlled trial will be conducted in a major paediatric hospital in Paris, France. Subjects will be divided into two arms. Each arm will contain 50 subjects.

For subjects of the Modeling arm, drug concentration will be measured at the 3rd hour of treatment and dosage adjustment will be done at the 6th hour of treatment using a bayesian approach. Vancomycin serum concentration will be then measured at the 24th hour of treatment.

Subjects of the control arm will receive the usual treatment strategy. Vancomycin serum concentration will be measured at the 24th hour of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 months to 16 years
* Children for whom a vancomycin treatment is started in the hospital Necker-Enfants Malades in Paris, France
* No objection of parents and of the child himself if he is able to express it.

Exclusion Criteria:

* Patients undergoing hemodialysis
* Patients undergoing peritoneal dialysis
* Newborns less than 1 months old
* Adolescents more than 16 years old and adults

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with vancomycin AUC/MIC ≥ 400 and serum trough concentration ≤ 20 mg/L | 24th hour of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TRELUYER, MD, PhD, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan DR, Anderson RL. A simple procedure for adjusting eyelid position after aponeurotic ptosis surgery. Arch Ophthalmol. 1987 Sep;105(9):1288-91. doi: 10.1001/archopht.1987.01060090146046. PMID 3632448
- [Background] Hikida RS, Lombardo JA. Regeneration of pigeon fast and slow muscle fiber types after partial excision and mincing. J Cell Biol. 1974 May;61(2):414-26. doi: 10.1083/jcb.61.2.414. PMID 4275137
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Result] Berthaud R, Benaboud S, Hirt D, Genuini M, Oualha M, Castelle M, Briand C, Artru S, Norsa L, Boyer O, Foissac F, Bouazza N, Treluyer JM. Early Bayesian Dose Adjustment of Vancomycin Continuous Infusion in Children: a Randomized Controlled Trial. Antimicrob Agents Chemother. 2019 Sep 9;63(12):e01102-19. doi: 10.1128/AAC.01102-19. Epub 2019 Oct 7. PMID 31591117